CLINICAL TRIAL: NCT00676052
Title: Multicentre Dose Ranging Study for Once Daily GSK233705 in COPD
Brief Title: Dose-Ranging Study Of GSK233705B In Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC2110664
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Results first posted 2017-09-07 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Multicenter; GSK233705B; double-blind; Chronic Obstructive Pulmonary Disease (COPD); randomized
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental): GSK233705 12.5mcg
  Interventions: Drug: GSK233705 12.5mcg
- Arm 2 (Experimental): GSK233705 25mcg
  Interventions: Drug: GSK233705 25mcg
- Arm 3 (Experimental): GSK233705 50mcg
  Interventions: Drug: GSK233705 50mcg
- Arm 4 (Experimental): GSK233705 100mcg
  Interventions: Drug: GSK233705 100mcg
- Arm 5 (Experimental): GSK233705 200mcg
  Interventions: Drug: GSK233705 200mcg
- Arm 6 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK233705 12.5mcg — Once daily via dry powder inhaler
  Arms: Arm 1
Drug: GSK233705 25mcg — once daily via dry powder inhaler
  Arms: Arm 2
Drug: GSK233705 50mcg — Once daily via dry powder inhaler
  Arms: Arm 3
Drug: GSK233705 100mcg — Once daily via dry powder inhaler
  Arms: Arm 4
Drug: GSK233705 200mcg — Once daily via dry powder inhaler
  Arms: Arm 5
Drug: Placebo — Once daily via dry powder imhaler
  Arms: Arm 6

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of GSK233705B compared with placebo in subjects with COPD.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated written informed consent prior to study participation.
* Male or female adults.

A female is eligible to enter and participate in this study if she is of:

non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who is post-menopausal; or child-bearing potential, has a negative pregnancy test at Visit 1/Visit 1A, and agrees to one of the protocol-specified acceptable contraceptive methods used consistently and correctly (i.e. according to the approved product label and the instructions of the physician for the duration of the study - Screening through follow-up contact)

* 40 to 80 years of age at Visit 1
* An established clinical history of COPD
* Current or previous cigarette smokers with a history of cigarette smoking of ≥ 10 pack-years 1.
* A post-albuterol/salbutamol FEV1/FVC ratio of ≤0.70 and a post-albuterol/salbutamol FEV1 of ≥35 and ≤70% of predicted normal values

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Women who are pregnant or lactating.
* A current diagnosis of asthma.
* Known respiratory disorders other than COPD including but not limited to α-1 antitrypsin deficiency as the underlying cause of COPD, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, and interstitial lung disease.
* Any previous lung resection surgery (e.g., lung volume reduction surgery or lobectomy)
* Clinically significant Chest X-ray or computed tomography (CT) scan abnormalities within 6 months prior to Visit 1 that are not believed to be due to COPD.
* Use of oral corticosteroids or antibiotics for COPD within 6 weeks prior to Visit 1.
* Hospitalization for COPD or pneumonia within 3 months prior to Visit 1.
* Use of antibiotics for a lower respiratory tract infection within 30 days prior to Visit 1.
* Clinically significant and uncontrolled cardiovascular, neurological, psychiatric, renal, gastro-intestinal, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities.
* An abnormal and clinically significant 12-lead electrocardiogram (ECG) that results in active medical problem.
* Positive for Hepatitis B or Hepatitis C at Visit 1.
* A current malignancy or previous history of cancer in remission for <5 years prior to Visit 1
* A history of allergy or hypersensitivity to ipratropium, tiotropium, or atropine and any of their derivatives, lactose/milk protein or magnesium stearate.
* Medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the study investigator would prevent use of an inhaled anticholingeric.
* Medically unable to withhold albuterol/salbutamol for 6 hours prior to spirometry testing at each study visit or to withhold ipratropium (if applicable) for the 6-hour period prior to the first 3 study visits (ipratropium cannot be used after Visit 3).
* Additional Medications: Unable to stop using certain medications such as bronchodilators and corticosteroids for the protocol-specified times prior to Visit 1 (the Investigator will discuss the specific medications)
* Use of inhaled corticosteroids at a dose greater than 1000 mcg/day of fluticasone propionate or equivalent within 30 days prior to Visit 1.
* Use of long-term oxygen therapy (LTOT) or supplemental oxygen required for greater than 12 hours a day. Oxygen use as needed is not exclusionary.
* Clinically significant sleep apnea that requires continuous positive airway pressure (CPAP)
* Use of regular nebulized therapy
* Use of nocturnal positive pressure or non-invasive positive pressure ventilation (NIPPV)
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1.
* An investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the above who is involved in this study
* History of psychiatric disease, intellectual deficiency, poor motivation, substance abuse in the two years prior to Visit 1 (including drug and alcohol), or other conditions, which will limit the validity of informed consent to participate in the study.
* Use of GSK233705B in previous studies.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2008-05-16 (Actual); Primary Completion 2008-12-22 (Actual); Study Completion 2008-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (75):
- United States (24):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Argentina (4):
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Pergamino, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán
- Bulgaria (3):
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
- Canada (8):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Sainte Jerome, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- Chile (3):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Germany (8):
  - GSK Investigational Site, Wiesloch, Baden-Wurttemberg
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
- Hungary (3):
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Mátraháza
- Netherlands (4):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Hoorn
- Philippines (2):
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, Quezon City
- Romania (3):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
- South Africa (5):
  - GSK Investigational Site, Cape Town, Gauteng
  - GSK Investigational Site, Mueckelneck, Gauteng
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Mowbray
- GSK Investigational Site, Seoul, South Korea
- Thailand (4):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Songkhla
- United Kingdom (3):
  - GSK Investigational Site, Brighton, Sussex East
  - GSK Investigational Site, London
  - GSK Investigational Site, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bateman E, Feldman G, Kilbride S, Brooks J, Mehta R, Harris S, Maden C, Crater G. Efficacy and safety of the long-acting muscarinic antagonist GSK233705 delivered once daily in patients with COPD. Clin Respir J. 2012 Oct;6(4):248-57. doi: 10.1111/j.1752-699X.2011.00278.x. Epub 2012 Feb 13. PMID 22329914
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: AC2110664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC2110664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC2110664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AC2110664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC2110664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AC2110664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC2110664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 79 centers: 30 in North America, 28 in Europe and 21 in International regions. The first participant first visit was on 16 May 2008 and last participant last visit was on 22 December 2008.
Pre-assignment Details: Out of the 963 participants screened for this study, 303 participants were screen failures and 79 participants were run-in failures. Therefore, a total of 581 participants were randomized out of which 5 participants did not receive any study medication, thus 576 participants were included in the intent-to-treat (ITT) Population.
Groups:
- Placebo: Eligible participants completed a two week run-in period during which they received placebo once daily via the novel dry powder inhaler. After run-in period, participants were randomized to receive placebo administered once daily via a novel dry powder inhaler.
- GSK233705B 12.5 mcg: Eligible participants completed a two week run-in period during which they received placebo once daily via the novel dry powder inhaler. After run-in period, participants were randomized to receive GSK233705B 12.5 micrograms (mcg) administered once daily via a novel dry powder inhaler.
- GSK233705B 25 mcg: Eligible participants completed a two week run-in period during which they received placebo once daily via the novel dry powder inhaler. After run-in period, participants were randomized to receive GSK233705B 25 mcg administered once daily via a novel dry powder inhaler.
- GSK233705B 50 mcg: Eligible participants completed a two week run-in period during which they received placebo once daily via the novel dry powder inhaler. After run-in period, participants were randomized to receive GSK233705B 50 mcg administered once daily via a novel dry powder inhaler.
- GSK233705B 100 mcg: Eligible participants completed a two week run-in period during which they received placebo once daily via the novel dry powder inhaler. After run-in period, participants were randomized to receive GSK233705B 100 mcg administered once daily via a novel dry powder inhaler.
- GSK233705B 200 mcg: Eligible participants completed a two week run-in period during which they received placebo once daily via the novel dry powder inhaler. After run-in period, participants were randomized to receive GSK233705B 200 mcg administered once daily via a novel dry powder inhaler.
Period: Overall Study
Arm/Group | Placebo | GSK233705B 12.5 mcg | GSK233705B 25 mcg | GSK233705B 50 mcg | GSK233705B 100 mcg | GSK233705B 200 mcg
Started | 96 | 95 | 96 | 97 | 95 | 97
Completed | 87 | 88 | 90 | 92 | 89 | 91
Not Completed | 9 | 7 | 6 | 5 | 6 | 6
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 2 | 2
Not completed — Lack of Efficacy | 2 | 2 | 1 | 1 | 2 | 1
Not completed — Protocol Violation | 5 | 3 | 2 | 2 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population comprised of all participants randomized to treatment who received at least one dose of study medication.
Groups:
- GSK233705B 12.5 mcg: Eligible participants completed a two week run-in period during which they received placebo once daily via the novel dry powder inhaler. After run-in period, participants were randomized to receive GSK233705B 12.5 mcg administered once daily via a novel dry powder inhaler.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK233705B 12.5 mcg | GSK233705B 25 mcg | GSK233705B 50 mcg | GSK233705B 100 mcg | GSK233705B 200 mcg | Total
Number analyzed (Participants) | 96 | 95 | 96 | 97 | 95 | 97 | 576
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (8.73) | 62.2 (9.75) | 62.2 (8.70) | 62.8 (6.99) | 61.7 (8.77) | 64.1 (8.30) | 62.4 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 34 | 43 | 45 | 33 | 34 | 235
  Male | 50 | 61 | 53 | 52 | 62 | 63 | 341
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 0 | 1 | 3
  Asian | 8 | 7 | 4 | 7 | 8 | 9 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 5 | 2 | 3 | 2 | 16
  White | 84 | 86 | 86 | 88 | 83 | 85 | 512
  More than one race | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Day 29
Description: The trough FEV1 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Day 28. The Baseline FEV1 is the mean of the two assessments made 30 minutes pre-dose and immediately pre-dose [time 0] on Day 1. Change from Baseline was calculated by subtracting the post-baseline assessment value from the Baseline value.
Time Frame: Baseline (pre-dose Day 1) and Day 29
Population: ITT Population. Last observation carried forward (LOCF) data has been presented.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | GSK233705B 12.5 mcg | GSK233705B 25 mcg | GSK233705B 50 mcg | GSK233705B 100 mcg | GSK233705B 200 mcg | Placebo
Number analyzed (Participants) | 94 | 94 | 97 | 94 | 96 | 94
Liter | 0.058 (0.0180) | 0.088 (0.0180) | 0.060 (0.0178) | 0.073 (0.0181) | 0.128 (0.0179) | -0.009 (0.0181)
Statistical Analysis 1: Comparison: GSK233705B 12.5 mcg vs Placebo; Test type: Superiority; p = 0.009, ANCOVA — Analysis performed using ANCOVA with covariates of Baseline, sex, age, smoking status, responsiveness stratum and treatment. Missing trough FEV1 data at Day 29 was imputed using LOCF; Mean Difference (Net) = 0.067, 95% CI 2-sided [0.017 to 0.117]
Statistical Analysis 2: Comparison: GSK233705B 25 mcg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.097, 95% CI 2-sided [0.047 to 0.147]
Statistical Analysis 3: Comparison: GSK233705B 50 mcg vs Placebo; Test type: Superiority; p = 0.007, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.069, 95% CI 2-sided [0.019 to 0.118]
Statistical Analysis 4: Comparison: GSK233705B 100 mcg vs Placebo; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.082, 95% CI 2-sided [0.032 to 0.132]
Statistical Analysis 5: Comparison: GSK233705B 200 mcg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.137, 95% CI 2-sided [0.086 to 0.187]

2. Secondary Outcome: Change From Baseline in Weighted Mean for 0 to 24 Hours Serial FEV1 on Day 1 to 2 and 28 to 29
Description: Weighted means serial FEV1 was derived by calculating the area under curve (AUC), and then dividing by the time interval over which the AUC was calculated. Baseline was defined at pre-dose Day 1. The weighted mean change from Baseline is the weighted mean minus Baseline. The AUC was calculated using the trapezoidal rule. For all post-dose observations, actual times that the spirometry measurements were conducted was used for the calculation. Pre-dose observations were counted as 0 hr observations - that is they had their time set to the time of dosing. The pre-dose value used for the calculation of the AUC was the mean of the two pre-dose observations (-30 and 0 min for Day 1 or 28). If one of these observations was missing, the remaining single pre-dose observation was used.
Time Frame: Baseline (pre-dose Day 1) and Days 1 to 2, Days 28 to 29
Population: ITT Population. Participants with analyzable data on the indicated time point have been presented.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | GSK233705B 12.5 mcg | GSK233705B 25 mcg | GSK233705B 50 mcg | GSK233705B 100 mcg | GSK233705B 200 mcg | Placebo
Number analyzed (Participants) | 94 | 95 | 97 | 94 | 97 | 94
Liter
  FEV1, Day 1: number analyzed (Participants) | 93 | 92 | 96 | 94 | 96 | 93
  FEV1, Day 1 | 0.085 (0.0146) | 0.086 (0.0146) | 0.102 (0.0143) | 0.132 (0.0146) | 0.155 (0.0144) | -0.021 (0.0146)
  FEV1, Day 28: number analyzed (Participants) | 88 | 89 | 90 | 89 | 91 | 86
  FEV1, Day 28 | 0.087 (0.0180) | 0.122 (0.0179) | 0.105 (0.0178) | 0.122 (0.0180) | 0.150 (0.0178) | -0.020 (0.0182)
Statistical Analysis 1: Comparison: GSK233705B 12.5 mcg vs Placebo; FEV1, Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — Analysis performed using repeated measures with covariates of Baseline, sex, age, smoking status, responsiveness stratum, Day (nominal), treatment and Day by treatment and Day by Baseline interactions; Mean Difference (Net) = 0.106, 95% CI 2-sided [0.065 to 0.146]
Statistical Analysis 2: Comparison: GSK233705B 25 mcg vs Placebo; FEV1, Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.107, 95% CI 2-sided [0.067 to 0.147]
Statistical Analysis 3: Comparison: GSK233705B 50 mcg vs Placebo; FEV1, Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.123, 95% CI 2-sided [0.083 to 0.163]
Statistical Analysis 4: Comparison: GSK233705B 100 mcg vs Placebo; FEV1, Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.152, 95% CI 2-sided [0.112 to 0.193]
Statistical Analysis 5: Comparison: GSK233705B 200 mcg vs Placebo; FEV1, Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.176, 95% CI 2-sided [0.135 to 0.216]
Statistical Analysis 6: Comparison: GSK233705B 12.5 mcg vs Placebo; FEV1, Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.106, 95% CI 2-sided [0.056 to 0.157]
Statistical Analysis 7: Comparison: GSK233705B 25 mcg vs Placebo; FEV, Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.142, 95% CI 2-sided [0.092 to 0.192]
Statistical Analysis 8: Comparison: GSK233705B 50 mcg vs Placebo; FEV1, Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.124, 95% CI 2-sided [0.074 to 0.174]
Statistical Analysis 9: Comparison: GSK233705B 100 mcg vs Placebo; FEV1, Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.142, 95% CI 2-sided [0.092 to 0.193]
Statistical Analysis 10: Comparison: GSK233705B 200 mcg vs Placebo; FEV1, Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.170, 95% CI 2-sided [0.120 to 0.220]

3. Secondary Outcome: Change From Baseline in Weighted Mean for 0 to 24 Hours Forced Vital Capacity (FVC) on Day 1 to 2 and 28 to 29
Description: Weighted means serial FVC was derived by calculating the AUC, and then dividing by the time interval over which the AUC was calculated. Baseline was defined at pre-dose Day 1. The weighted mean change from Baseline is the weighted mean minus Baseline. The AUC was calculated using the trapezoidal rule. For all post-dose observations, actual times that the spirometry measurements were conducted was used for the calculation. Pre-dose observations were counted as 0 hr observations - that is they had their time set to the time of dosing. The pre-dose value used for the calculation of the AUC was the mean of the two pre-dose observations (-30 and 0 min for Day 1 or 28). If one of these observations was missing, the remaining single pre-dose observation was used.
Time Frame: Baseline (pre-dose Day 1) and Days 1 to 2, Days 28 to 29
Population: ITT Population. Participants with analyzable data on the indicated time point have been presented.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | GSK233705B 12.5 mcg | GSK233705B 25 mcg | GSK233705B 50 mcg | GSK233705B 100 mcg | GSK233705B 200 mcg | Placebo
Number analyzed (Participants) | 94 | 95 | 97 | 94 | 97 | 94
Liter
  Day 1: number analyzed (Participants) | 93 | 92 | 96 | 94 | 96 | 93
  Day 1 | 0.129 (0.0257) | 0.149 (0.0257) | 0.160 (0.0253) | 0.207 (0.0257) | 0.263 (0.0257) | -0.037 (0.0257)
  Day 28: number analyzed (Participants) | 88 | 89 | 90 | 89 | 91 | 86
  Day 28 | 0.137 (0.0287) | 0.178 (0.0285) | 0.150 (0.0283) | 0.191 (0.0287) | 0.253 (0.0283) | -0.041 (0.0289)
Statistical Analysis 1: Comparison: GSK233705B 12.5 mcg vs Placebo; Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.166, 95% CI 2-sided [0.094 to 0.237]
Statistical Analysis 2: Comparison: GSK233705B 25 mcg vs Placebo; Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.186, 95% CI 2-sided [0.115 to 0.258]
Statistical Analysis 3: Comparison: GSK233705B 50 mcg vs Placebo; Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.198, 95% CI 2-sided [0.127 to 0.268]
Statistical Analysis 4: Comparison: GSK233705B 100 mcg vs Placebo; Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.244, 95% CI 2-sided [0.172 to 0.315]
Statistical Analysis 5: Comparison: GSK233705B 200 mcg vs Placebo; Day 1; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.301, 95% CI 2-sided [0.229 to 0.372]
Statistical Analysis 6: Comparison: GSK233705B 12.5 mcg vs Placebo; Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.178, 95% CI 2-sided [0.098 to 0.258]
Statistical Analysis 7: Comparison: GSK233705B 25 mcg vs Placebo; Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.219, 95% CI 2-sided [0.139 to 0.298]
Statistical Analysis 8: Comparison: GSK233705B 50 mcg vs Placebo; Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.191, 95% CI 2-sided [0.111 to 0.270]
Statistical Analysis 9: Comparison: GSK233705B 100 mcg vs Placebo; Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.232, 95% CI 2-sided [0.152 to 0.312]
Statistical Analysis 10: Comparison: GSK233705B 200 mcg vs Placebo; Day 28; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.294, 95% CI 2-sided [0.214 to 0.373]

4. Secondary Outcome: Change From Baseline in Clinic Visit Trough FVC on Day 29
Description: The trough FVC is defined as the mean of the FVC values obtained 23 and 24 hours after dosing on Day 28. The Baseline FVC is the mean of the two assessments made 30 minutes pre-dose and immediately pre-dose [time 0] on Day 1. Change from Baseline was calculated by subtracting the post-baseline assessment value from the Baseline value.
Time Frame: Baseline (pre-dose Day 1) and Day 29
Population: ITT Population. Participants with analyzable data on the indicated time point have been presented.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | GSK233705B 12.5 mcg | GSK233705B 25 mcg | GSK233705B 50 mcg | GSK233705B 100 mcg | GSK233705B 200 mcg | Placebo
Number analyzed (Participants) | 88 | 90 | 91 | 89 | 91 | 87
Liter | 0.088 (0.0301) | 0.139 (0.0298) | 0.083 (0.0295) | 0.152 (0.0300) | 0.224 (0.0297) | -0.011 (0.0301)
Statistical Analysis 1: Comparison: GSK233705B 12.5 mcg vs Placebo; Test type: Superiority; p = 0.021, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.099, 95% CI 2-sided [0.015 to 0.182]
Statistical Analysis 2: Comparison: GSK233705B 25 mcg vs Placebo; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.150, 95% CI 2-sided [0.067 to 0.233]
Statistical Analysis 3: Comparison: GSK233705B 50 mcg vs Placebo; Test type: Superiority; p = 0.026, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.094, 95% CI 2-sided [0.011 to 0.177]
Statistical Analysis 4: Comparison: GSK233705B 100 mcg vs Placebo; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.163, 95% CI 2-sided [0.080 to 0.247]
Statistical Analysis 5: Comparison: GSK233705B 200 mcg vs Placebo; Test type: Superiority; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.235, 95% CI 2-sided [0.152 to 0.319]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected up to follow visit (7 to 9 days post visit 8 or premature discontinuation).
Description: ITT Population was used in the analysis of safety data.
Arm/Group | Placebo | GSK233705B 12.5 mcg | GSK233705B 25 mcg | GSK233705B 50 mcg | GSK233705B 100 mcg | GSK233705B 200 mcg
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/95 | 0/96 | 0/97 | 0/95 | 1/97
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/95 | 2/96 | 1/97 | 1/95 | 1/97
Other Adverse Events (participants affected / at risk) | 7/96 | 4/95 | 6/96 | 9/97 | 5/95 | 3/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=96) | GSK233705B 12.5 mcg (N=95) | GSK233705B 25 mcg (N=96) | GSK233705B 50 mcg (N=97) | GSK233705B 100 mcg (N=95) | GSK233705B 200 mcg (N=97)
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=96) | GSK233705B 12.5 mcg (N=95) | GSK233705B 25 mcg (N=96) | GSK233705B 50 mcg (N=97) | GSK233705B 100 mcg (N=95) | GSK233705B 200 mcg (N=97)
Headache (Nervous system disorders) | 7 (9) | 4 (4) | 6 (6) | 9 (14) | 5 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.